CLINICAL TRIAL: NCT03421860
Title: Cardiac Index Changes With Ephedrine, Phenylephrine, Ondansetron and Norepinephrine During Spinal Anesthesia for Cesarian Section
Brief Title: Cardiac Index Changes With Ephedrine, Phenylephrine, Ondansetron and Norepinephrine During Spinal Anesthesia
Acronym: EPhON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben marzouk Sofiene, MD, assistant professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: bich-fel
Record Dates: First submitted 2017-08-04; First posted 2018-02-05 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Cardiac Output, Low
Keywords: Spinal anesthesia; cardiac output; vasopressor
MeSH Terms: conditions — Cardiac Output, Low | interventions — Ephedrine; Cardiac Output; Phenylephrine; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ephedrine (Active Comparator): will receive ephedrine :a bolus of 9 mg after SA once intervention: will receive complementary doses of ephedrine 6 mgto maintain systolic blood pressure above 80 % of baseline
  Interventions: Drug: cardiac output changes with "ephedrine"
- phenylephrine (Active Comparator): will receive Phenylephrine : a bolus of 100 mcg once intervention: will receive complementary doses of ephedrine 6 mg to maintain systolic blood pressure above 80 % of baseline
  Interventions: Drug: cardiac output changes with "phenylephrine"
- ondansetron (Active Comparator): will receive ondansetron: a bolus of 8 mg once intervention: will receive complementary doses of ephedrine 6 mg to maintain systolic blood pressure above 80 % of baseline
  Interventions: Drug: cardiac output changes with "ondansetron"
- norepinephrine (Active Comparator): will receive noradrenaline (norepinephrine) a bolus of 0,25 mcg/kg once intervention: will receive complementary doses of ephedrine 6 mg to maintain systolic blood pressure above 80 % of baseline
  Interventions: Drug: cardiac output changes with "nor-epinephrine"

INTERVENTIONS:
Drug: cardiac output changes with "ephedrine" — measure cardiac output after giving a bolus of ephedrine intervention: will receive complementary doses of ephedrine to maintain systolic blood pressure above 80 % of baseline
  Other Names: cardiac output: CO (cm3 / min) = ITV * S * HR . ITV (cm) = integral time velocity is measured by pulsed doppler at the level of the ascending aorta, on apical cut.
  Arms: ephedrine
Drug: cardiac output changes with "phenylephrine" — measure cardiac output after giving a bolus of phenylephrine intervention: will receive complementary doses of ephedrine to maintain systolic blood pressure above 80 % of baseline
  Other Names: cardiac output: CO (cm3 / min) = ITV * S * HR. ITV (cm) = integral time velocity is measured by pulsed doppler at the level of the ascending aorta, on apical cut.
  Arms: phenylephrine
Drug: cardiac output changes with "ondansetron" — measure cardiac output after giving a bolus of ondansetron intervention: will receive complementary doses of ephedrine to maintain systolic blood pressure above 80 % of baseline
  Other Names: cardiac output: CO (cm3 / min) = ITV * S * HR. ITV (cm) = integral time velocity is measured by pulsed doppler at the level of the ascending aorta, on apical cut.
  Arms: ondansetron
Drug: cardiac output changes with "nor-epinephrine" — measure cardiac output after giving a bolus of nor-epinephrine intervention: will receive complementary doses of ephedrine to maintain systolic blood pressure above 80 % of baseline
  Other Names: cardiac output: CO (cm3 / min) = ITV * S * HR. ITV (cm) = integral time velocity is measured by pulsed doppler at the level of the ascending aorta, on apical cut.
  Arms: norepinephrine

SUMMARY:
The purpose of the study is to evaluate the cardiac output changes after an intravenous bolus of ephedrine, phenylephrine, ondansetron or norepinephrine during a spinal anesthetic for a cesarean delivery.

For elective cesarean delivery, all participants will receive spinal anesthesia with a local anesthetic and sufentanil. This study includes 120 pregnant women. Patients will be randomly assigned according to a computer generated system to be in one of four groups.

DETAILED DESCRIPTION:
This study will be a prospective, randomized, double-blind controlled trial. After written and informed consent are obtained, the study participants are randomly assigned using a computer generated table to 1 of 4 treatment groups prior to cesarean delivery.

Group A: 9 mg of ephedrine Group B: 100 mcg of phenylephrine Group C: 8 mg of ondansetron Group D: 0,25 mcg/kg of norepinephrine Baseline arterial blood pressure and heart rate will be measured in the left lateral tilt position, before anesthesia and then every minute.The cardiac output is calculated on the apical cut 5 cavities, before anesthesia and then every 5 miutes. No fluid preloading will be administered till delivery.

The primary endpoint is cardiac output changes in each groups. The secondary endpoint is the number of provider interventions needed to maintain the SBP within 80-120% of baseline for each groups.

Bradycardia (HR less than 50 BPM) will be treated with 1 mg of Atropine. Hypotension ( decrease of more than 20% of the baseline value or a PAS <90 mm Hg) will be treated with 6 mg of ephedrine, without any fluid loading.

The spinal anesthesia will be carried out in a seated position, level L3-L4 or L4-L5 with a slow injection over 30 seconds of a mixture of 10 mg of 0.5% Bupivacaine with 5 mcg of Sufentanil. The hot / cold test to determine the block level is required. A spinal anesthesia is validated if the cold test reaches the T4 level. The 10 ml syringe will be administered immediately after spinal anesthesia. The patient will be placed in the left lateral tilt position of 15¤, then put back into strict DD immediately after the delivery. Cardiovascular parameters (PAS, PAM, PAD, HR) will be recorded every minute until delivery. Echocardiographic measurement of cardiac output will be recorded every five minutes until delivery.

Measured variables will include systolic, diastolic and mean non-invasive blood pressure, the number and type of interventions for control of blood pressure, heart rate, cardiac output, incidence of nausea and vomiting (NV), incidence of arrhythmia and fetal cord blood analysis (pH) at delivery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I / II
* Caesarean section, non-twinned

Exclusion Criteria:

* heart disease
* HTA
* non-gestational diabetes
* pre-eclampsia
* sepsis
* BMI greater than 40
* contraindication to spinal anesthesia: patient refusal, medicinal allergy, long QT syndrome.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
cardiac output changes for 120 patients | at time of delivery (right after spinal anesthesia until delivery)
  In left lateral tilt position, cardiac output is calculated on the echocardiographic apical cut 5 cavities, every 5 minutes till delivery, with an infusion of either Ephedrine, Phenylephrine, Ondansetron or Norepinephrine.
  The cardiac output is calculated on the apical cut 5 cavities:
  Dc (cm3 / min) = ITV * S * HR Dc = cardiac output ITV (cm) = integral time velocity is measured by pulsed doppler at the level of the ascending aorta, on apical cut. Only the closing click (B2) is visible.
  If B2 is not visible, the sample is placed too much in the hunting chamber, which underestimates the ITV.
  If B1 and B2 are visible, the sample is too close to the aortic ring, which overestimates the ITV measurement.
  S = surface area of the aortic ring = (aorta diameter) ₂ * π / 4 The diameter of the aorta is the average of three measurements at the beginning of systole, on the major axis.

SECONDARY OUTCOMES:
Maternal Blood Pressure | at time of delivery (right after spinal anesthesia until delivery)
  Measurement of systolic, diastolic and mean, non-invasive blood pressure during cesarean delivery with an infusion of either Ephedrine, Phenylephrine, Ondansetron or Norepinephrine
heart rate | at time of delivery (right after spinal anesthesia until delivery)
  mean heart rate during cesarean delivery with an infusion of either Ephedrine, Phenylephrine, Ondansetron or Norepinephrine
Vomiting | at time of delivery (right after spinal anesthesia until delivery)
  incidence of Vomiting during cesarean section with an infusion of either Ephedrine, Phenylephrine, Ondansetron or Norepinephrine
mean pH of the fetal cord blood | at time of delivery (right after spinal anesthesia until delivery)
  fetal cord blood analysis will be done immediately after delivery in order to determine the pH value in each group
Nausea | at time of delivery (right after spinal anesthesia until delivery)
  incidence of nausea during cesarean section with an infusion of either Ephedrine, Phenylephrine, Ondansetron or Norepinephrine

CONTACTS AND LOCATIONS:
Overall Officials: hayen maghrebi, professor, Study Chair — tunis maternity center
Locations (1):
- Tunis maternity and neonatology center, minisetry of public health, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No